CLINICAL TRIAL: NCT00187096
Title: Pilot Study Of Haplo-Identical Natural Killer Cell Transplantation For Acute Myeloid Leukemia
Brief Title: Natural Killer (NK) Cell Transplantation for AML
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NKAML
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2012-11-09 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2013-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: Leukemia; Myeloid; Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — Cyclophosphamide; fludarabine; Clofarabine; Etoposide; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stratum 1 (Experimental): Stratum 1 (AML in complete remission)
  Cyclophosphamide 60 mg/kg IV Day -7 Fludarabine 25 mg/m2/day IV Days -6 through -2 Donor pheresis Day -1 Start IL-2 on Day -1, then 3 times per week x 2 weeks NK Cell purification and infusion on Day 0
  Interventions: Drug: Cyclophosphamide, Fludarabine, Clofarabine, Etoposide, Interleukin-2; Procedure: Natural Killer Cell Infusion; Device: CliniMACS System
- Stratum 2 (Experimental): Stratum 2 (AML that is refractory or relapsed or AML with increasing minimal residual disease)
  Clofarabine 40 mg/m2 IV, days -6 through -2 Etoposide 100 mg/m2 IV, days -6 through -2 Cyclophosphamide 400 mg/m2 IV, days -6 through 02 Donor pheresis Day -1 Start IL-2 Day -1, and then 3 times per week x 2 weeks NK Cell purification and infusion on Day 0.
  Interventions: Drug: Cyclophosphamide, Fludarabine, Clofarabine, Etoposide, Interleukin-2; Procedure: Natural Killer Cell Infusion; Device: CliniMACS System

INTERVENTIONS:
Drug: Cyclophosphamide, Fludarabine, Clofarabine, Etoposide, Interleukin-2 — See Detailed Description section for additional details of treatment interventions.
Procedure: Natural Killer Cell Infusion — See Detailed Description section for additional details of treatment interventions.
Device: CliniMACS System — See Detailed Description section for additional details of treatment interventions.

SUMMARY:
The purpose of this study is to assess the safety and efficacy of infusing natural killer cells from a donor as treatment for patients with acute myeloid leukemia in remission or who have experienced relapse.

DETAILED DESCRIPTION:
Natural killer (NK) cells extracted from a [parental] donor are infused intravenously. Most patients are given a multi-agent chemotherapeutic conditioning regimen prior to the infusion. The conditioning regimen may be omitted for patients who have previously received traditional stem cell transplant.

Details of Treatment Plan:

Stratum 1 (AML in complete remission)

Cyclophosphamide 60 mg/kg IV Day -7 Fludarabine 25 mg/m2/day IV Days -6 through -2 Donor pheresis Day -1 Start IL-2 on Day -1, then 3 times per week x 2 weeks NK Cell purification and infusion on Day 0

Stratum 2 (AML that is refractory or relapsed or AML with increasing minimal residual disease)

Clofarabine 40 mg/m2 IV, days -6 through -2 Etoposide 100 mg/m2 IV, days -6 through -2 Cyclophosphamide 400 mg/m2 IV, days -6 through 02 Donor pheresis Day -1 Start IL-2 Day -1, and then 3 times per week x 2 weeks NK Cell purification and infusion on Day 0.

For patients who have received prior SCT, the conditioning regimen may be omitted if the NK cells are obtained from the original SCT donor.

Cytokine regimen (stratum 1 and 2): 1 million units/m2 of IL-2 given subcutaneously three times per week for two weeks (6 doses) starting on the evening of day -1.

NK Cell Transplantation (stratum 1 and 2): NK cells from haplo-identical family donor will be infused on day 0.

ELIGIBILITY:
Inclusion Criteria:

* Participants with AML that is in complete remission, is relapsed or refractory, or with increasing minimal residual disease.
* Participants in complete remission must have recovered from toxicity of previous therapy and have evidence of bone marrow recovery
* Participants who had prior stem cell transplant (SCT) must have no evidence of GVHD and 60 or more days have elapsed since the SCT.

Exclusion Criteria:

* Participants who are pregnant
* Participants with inadequate renal, liver, or pulmonary functions

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2005-09; Primary Completion 2012-02 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey E. Rubnitz, M.D., Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Result] Rubnitz JE, Inaba H, Ribeiro RC, Pounds S, Rooney B, Bell T, Pui CH, Leung W. NKAML: a pilot study to determine the safety and feasibility of haploidentical natural killer cell transplantation in childhood acute myeloid leukemia. J Clin Oncol. 2010 Feb 20;28(6):955-9. doi: 10.1200/JCO.2009.24.4590. Epub 2010 Jan 19. PMID 20085940
- See also: St. Jude Children's Research Hospital — http://www.stjude.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 49 participants were recruited between October 2005 and October 2011.
Pre-assignment Details: 49 participants were enrolled on the study. This report is based on results for 25 patients. 24 were donors and were excluded. All analyses are based on the intent-to-treat principle and therefore include all recipients with data available for the reported endpoint.
Groups:
- Arm 1: Conditioning Regimen: Cyclophosphamide/Fludarabine: Participants with AML in complete remission (stratum 1). AML in complete remission is defined as trilineage hematopoietic recovery with less than 5% blasts in the marrow. Arm 1 participants received a traditional conditioning regimen of cyclophosphamide and fludarabine prior to NK cell transplantation.
- Arm 2a: Conditioning Regimen: Cyclophosphamide/Fludarabine: AML that is refractory or relapsed or AML with increasing minimal residual disease (MRD) (stratum 2). Participants enrolled prior to Amendment 2.0 received a traditional conditioning regimen of cyclophosphamide and fludarabine prior to NK cell transplantation.
- Arm 2b: Conditioning: Clofarabine/Etoposide/Cyclophosphamide: AML that is refractory or relapsed or AML with increasing minimal residual disease (MRD) (stratum 2). Participants enrolled after protocol Amendment 2.0 received a novel conditioning regimen of clofarabine, etoposide and cyclophosphamide prior to NK cell transplantation.
Period: Overall Study
Arm/Group | Arm 1: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2a: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2b: Conditioning: Clofarabine/Etoposide/Cyclophosphamide
Started | 10 | 3 | 12
Completed | 10 | 3 | 11
Not Completed | 0 | 0 | 1
Not completed — unacceptable toxicity | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Conditioning Regimen: Cyclophosphamide/Fludarabine: AML in complete remission (stratum 1). AML in complete remission is defined as trilineage hematopoietic recovery with less than 5% blasts in the marrow. Arm 1 participants received a traditional conditioning regimen of cyclophosphamide and fludarabine prior to NK cell transplantation.
- Total: Total of all reporting groups
Arm/Group | Arm 1: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2a: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2b: Conditioning: Clofarabine/Etoposide/Cyclophosphamide | Total
Number analyzed (Participants) | 10 | 3 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.26 (7.74) | 6.05 (6.46) | 10.11 (5.9) | 8.48 (6.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 4 | 9
  Male | 5 | 3 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Experiencing Grade 3 or 4 Toxicities During Conditioning and up to 100 Days Post-transplant
Description: Document the number of patients experiencing grade 3 or 4 toxicities during conditioning and up to 100 days post-transplant. Toxicities were identified using Common Toxicity Criteria V 3.0 criteria.
Time Frame: Beginning at on therapy through 100 days post-transplant
Population: Grade 3 and 4 toxicities were assessed using Common Toxicity Criteria V.3.0 The assessment period was from the date on therapy through 100 days post-transplant.
Measure: Number; unit: participants
Groups:
- Arm 1: Conditioning Regimen: Cyclophosphamide/Fludarabine: AML in complete remission (stratum 1). AML in complete remission is defined as trilineage hematopoietic recovery with less than 5% blasts in the marrow. Participants received a traditional conditioning regimen of cyclophosphamide and fludarabine prior to NK cell transplantation.
- Arm 2a: Conditioning Regimen: Cyclophosphamide/Fludarabine: AML that is refractory or relapsed or AML with increasing minimal residual disease (MRD). Participants enrolled prior to Amendment 2.0 received a traditional conditioning regimen of cyclophosphamide and fludarabine prior to NK cell transplantation.
  Refractory: ≥ 20% leukemic blasts in the bone marrow or no decrease in the percentage of blasts in the bone marrow (e.g., if a patient starts with 15% blasts and still has 15% blasts, he would have refractory disease).
  Relapse: presence of ≥ 20% leukemic blasts in the bone marrow or the development of extramedullary disease after CR is achieved.
  Increasing Minimal Residual Disease (MRD) indicates higher MRD levels.
- Arm 2b: Conditioning: Clofarabine/Etoposide/Cyclophosphamide: AML that is refractory or relapsed or AML with increasing minimal residual disease (MRD) (stratum 2). Participants enrolled after protocol Amendment 2 received a novel conditioning regimen of clofarabine, etoposide and cyclophosphamide prior to NK cell transplantation.
Arm/Group | Arm 1: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2a: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2b: Conditioning: Clofarabine/Etoposide/Cyclophosphamide
Number analyzed (Participants) | 10 | 3 | 12
participants | 2 | 3 | 11

2. Primary Outcome: Proportion of Patients Experiencing Grade 3 or 4 Toxicities During Conditioning and up to 100 Days Post-transplant
Description: Document the proportion of patients experiencing grade 3 or 4 toxicities during conditioning and up to 100 days post-transplant. Toxicities were identified using Common Toxicity Criteria V 3.0 criteria.
Time Frame: Beginning at on therapy through 100 days post-transplant
Population: as for outcome 1
Measure: Number; unit: proportion of patients
Arm/Group | Arm 1: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2a: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2b: Conditioning: Clofarabine/Etoposide/Cyclophosphamide
Number analyzed (Participants) | 10 | 3 | 12
proportion of patients | 0.20 | 1.00 | 0.917

3. Secondary Outcome: Duration of Engraftment of Natural Killer (NK) Cells
Description: NK cell engraftment defined as NK cell chimerism in recipients.
Time Frame: Measured at days 2, 7, 14, 21 and 28 after NK cell transplantation, and up to 189 days post transplant as clinically indicated
Population: Arm 2 participants were not analyzed for this outcome as many of these patients proceeded to allogeneic stem cell transplantation following NK cell transplantation.
Measure: Median (Full Range); unit: Days
Arm/Group | Arm 1: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2a: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2b: Conditioning: Clofarabine/Etoposide/Cyclophosphamide
Number analyzed (Participants) | 10 | 0 | 0
Days | 10 [2 to 189] |  |

4. Secondary Outcome: Percent of Peak NK Cell Chimerism
Description: The maximum percent of donor NK cell in recipients during a four-week period after NK cell infusion.
Time Frame: Days 2, 7, 14, 21 and 28 after NK cell transplantation
Population: as for outcome 3
Measure: Median (Full Range); unit: percent of NK cells
Arm/Group | Arm 1: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2a: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2b: Conditioning: Clofarabine/Etoposide/Cyclophosphamide
Number analyzed (Participants) | 10 | 0 | 0
percent of NK cells | 7 [1 to 30] |  |

5. Secondary Outcome: Percent of Detectable Donor NK Cells at Day 28
Description: The percent of detectable donor NK cells in recipients at 28 days after NK cell infusion. Three of 10 participants had detectable donor cells at week 4. The results report the percent of detectable cells in the 3 participants.
Time Frame: At 28 days
Population: Three of 10 participants continued to have detectable donor NK cells at week 4.
Measure: Median (Full Range); unit: percent of donor NK cells
Arm/Group | Arm 1: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2a: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2b: Conditioning: Clofarabine/Etoposide/Cyclophosphamide
Number analyzed (Participants) | 3 | 0 | 0
percent of donor NK cells | 29 [7 to 30] |  |

6. Secondary Outcome: Day That Maximum NK Cell Engraftment Was Reached
Description: The time elapsed after transplantation in days until peak KIR-mismatched donor NK cell expansion was reached in recipients
Time Frame: Day 0 through Day 28 post NK cell transplantation
Population: Nine of the 10 participants in Arm 1 received KIR-mismatched NK donor cells.
Measure: Median (Full Range); unit: number of days
Arm/Group | Arm 1: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2a: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2b: Conditioning: Clofarabine/Etoposide/Cyclophosphamide
Number analyzed (Participants) | 9 | 0 | 0
number of days | 14 [7 to 28] |  |

7. Secondary Outcome: Number of KIR-mismatched NK Cells
Description: Number of KIR-mismatched donor NK cells in recipients' blood at day 2 and day 14 post NK cell infusion.
Time Frame: Day 2 and day 14 post NK cell transplantation
Population: Nine of the 10 participants in Arm 1 received KIR-mismatched NK donor cells.
Measure: Median (Full Range); unit: cells/µl
Arm/Group | Arm 1: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2a: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2b: Conditioning: Clofarabine/Etoposide/Cyclophosphamide
Number analyzed (Participants) | 9 | 0 | 0
cells/µl
  Day 2 | 210 [0 to 740] |  |
  Day 14 | 5,800 [220 to 27,400] |  |

8. Secondary Outcome: Number of Participants With Evidence of NK Cells Lysing a Target Cell Line (K562)
Description: NK cells in recipient achieving ability to lyse target cell line (K562) within normal range established by donor NK cells.
Time Frame: Days 2, 7, 14, 21, and 28 after NK cell transplantation
Population: All 10 participants received NK donor cells; 9 of the 10 participants received KIR-mismatched NK donor cells.
Measure: Number; unit: participants
Arm/Group | Arm 1: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2a: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2b: Conditioning: Clofarabine/Etoposide/Cyclophosphamide
Number analyzed (Participants) | 10 | 0 | 0
participants
  Lysed within normal range | 10 |  |
  Did not Lyse within normal range | 0 |  |

9. Secondary Outcome: Relapse-free Survival
Description: For Arm 1, the efficacy of NK cell transplantation will be reported as the proportion of participants who achieve complete or partial remission. Kaplan-Meier estimates of relapse-free survival and confidence interval was determined by binomial distribution because no events were observed. The binomial interval is based on the number of patients at risk.
Time Frame: Up to 2 years post NK cell transplantation
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Arm 1: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2a: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2b: Conditioning: Clofarabine/Etoposide/Cyclophosphamide
Number analyzed (Participants) | 10 | 0 | 0
Percent probability | 100 (0) [65.5 to 100] |  |

10. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time relapse from on study date to death with those alive at last follow up date censored. The Kaplan-Meier method was used to compute survival probability estimates and confidence interval was determined by binomial distribution (for no events or all events) or by log hazard method. The binomial interval is based on the number of patients at risk.
  The confidence intervals for Arm 1 and Arm 2a were determined by binomial distribution.
  The confidence interval for Arm 2b was determined by log hazard method.
Time Frame: Up to 2 years post NK cell transplantation
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Arm 1: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2a: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2b: Conditioning: Clofarabine/Etoposide/Cyclophosphamide
Number analyzed (Participants) | 10 | 3 | 12
Percent probability | 100 (0) [65.5 to 100] | 0 (0) [0 to 69] | 45.0 (13.6) [15.5 to 71.0]

ADVERSE EVENTS:
Time Frame: Beginning at on therapy through 100 days post-transplant
Arm/Group | Arm 1: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2a: Conditioning Regimen: Cyclophosphamide/Fludarabine | Arm 2b: Conditioning: Clofarabine/Etoposide/Cyclophosphamide
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/3 | 2/12
Other Adverse Events (participants affected / at risk) | 1/10 | 3/3 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Conditioning Regimen: Cyclophosphamide/Fludarabine (N=10) | Arm 2a: Conditioning Regimen: Cyclophosphamide/Fludarabine (N=3) | Arm 2b: Conditioning: Clofarabine/Etoposide/Cyclophosphamide (N=12)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatobiliary/Pancreas - Other (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils, blood (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils, Rectum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Conditioning Regimen: Cyclophosphamide/Fludarabine (N=10) | Arm 2a: Conditioning Regimen: Cyclophosphamide/Fludarabine (N=3) | Arm 2b: Conditioning: Clofarabine/Etoposide/Cyclophosphamide (N=12)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Typhlitis (cecal inflammation) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage, GI, Oral cavity (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage, pulmonary/upper respiratory, Nose (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage/Bleeding - Other (Specify, __) (General disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia-fever of unknown origin without clinically or microbiologically documented infe (Infections and infestations) | 1 (1) | 1 (1) | 5 (9)
Infection - Other (Specify, __) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils, Blood (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
Infection with normal ANC or Grade 1 or 2 neutrophils, Blood (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Phosphate, serum-low (hypokalemia) (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (3)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils, Lip/perioral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils, Rectum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes